CLINICAL TRIAL: NCT03988894
Title: Design, Usability Testing, and Feasibility Testing of a Smartphone App (mDASHNa-CC) to Support Healthy Diet and Hypertension Control for Chinese Canadian Seniors
Brief Title: mDASHNa-CC APP to Support a Healthy Diet and Hypertension Control for Chinese Canadian Seniors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Ping Zou, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02579746
Record Dates: First submitted 2019-06-08; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Diet, Healthy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: A pilot two-group (1:1) randomized controlled trial with a sample size of 60 (block of 20) in a Chinese Canadian community in the Greater Toronto Area, Ontario, Canada.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Usual Care (No Intervention): All participants will (a) receive a general hypertension health education booklet from the Heart and Stroke Foundation of Ontario;(b) be encouraged to see their family physicians or primary health care providers regarding their blood pressure status; those who do not have a primary health care provider will be referred to a walk-in clinic or a community health centre; and (c) have access to family physicians, tele-health, emergency care, hospital and other health care facilities in the Greater Toronto Area as required.
- Intervention: mDASHNa-CC app use (Active Comparator): In addition to usual care, those participants randomized to the intervention group will be offered use of the app.Then, they will load the app in their smartphones and be requested to review educational contents, conduct dietary self-assessment, and monitor blood pressure for 8 weeks.By the end of eight weeks post randomization, seniors will be prompted by phone using an audible alert to complete the app Evaluation Questionnaire on the smartphone, which ascertains likes and dislikes with the app.
  Interventions: Device: mDASHNa App

INTERVENTIONS:
Device: mDASHNa App — The functions of the app will include: (a) antihypertensive dietary education; (b) dietary self-assessment; (c) automatic feedback according to dietary self-assessment; (d) blood pressure monitoring; and (e) automatic feedback according to blood pressure data.
  Arms: Intervention: mDASHNa-CC app use

SUMMARY:
The aim of this proposed study is to translate the Dietary Approach to Stop Hypertension with Sodium (Na) Reduction for Chinese Canadian (DASHNa-CC), a classroom-based antihypertensive dietary educational intervention, to an innovative smartphone app (mDASHNa-CC) to enable Chinese Canadian seniors' access to this antihypertensive dietary intervention anytime, regardless of where they are.

ELIGIBILITY:
Inclusion Criteria:

* have a systolic blood pressure higher than 140 mmHg, or a diastolic blood pressure higher than 90mmHg, or are on antihypertensive medications, based on pre-intervention baseline assessment
* are able to understand (listen) and speak in Mandarin or Cantonese, read and write in Chinese
* have access to a smartphone

Exclusion Criteria:

* have special dietary requirements
* are a household member of another mDASHNa-CC participant
* plan to leave the area prior to the anticipated end of study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
change of systolic Blood Pressure from baseline to eight weeks after randomization | eight weeks after randomization
  Systolic blood pressures will be measured by the home blood pressure monitor, Omron BP785, whose validity and reliability have been tested
change of diastolic Blood Pressure from baseline to eight weeks after randomization | eight weeks after randomization
  diastolic blood pressures will be measured by the home blood pressure monitor, Omron BP785, whose validity and reliability have been tested
change of body weight from baseline to eight weeks after randomization | eight weeks after randomization
  Weight will be measured by an electronic body weight scale (Rubbermaid® Digital Utility Scale, Model number H-479, Capacity/Accuracy 400 lbs * 0.5 lb)
change of waist circumference from baseline to eight weeks after randomization | eight weeks after randomization
  Waist circumference will be measured by measurement tape following proper technique
change of Health-related Quality of Life from baseline to eight weeks after randomization | eight weeks after randomization
  Health-related quality of life will be measured by Medical Outcomes Study 36-Item Short Form version two. The SF-36v2 required ten minutes to complete and consisted of 36 items and eight domains, which could be grouped into physical and mental component summaries. All domains were scored on a scale ranging from 0 to 100, wherein 0 represented the worst overall health status and 100 the best health status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zou P, Stinson J, Parry M, Dennis CL, Yang Y, Lu Z. A Smartphone App (mDASHNa-CC) to Support Healthy Diet and Hypertension Control for Chinese Canadian Seniors: Protocol for Design, Usability and Feasibility Testing. JMIR Res Protoc. 2020 Apr 2;9(4):e15545. doi: 10.2196/15545. PMID 32238343